CLINICAL TRIAL: NCT05782439
Title: Detection of the Ileotibial Band Tension Through Direct Palpation: a Reliability Assessment Study
Brief Title: Palpation of the Ileotibial Band Tension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manusapiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ITB01
Record Dates: First submitted 2023-02-16; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: ileotibial band; clinical-test; direct palpation

STUDY DESIGN:
Intervention Model Description: Three different group (40, 20 and 40 subjects respectively) are enrolled in sequence and undergo the same evaluation procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adults (Experimental): Manual and instrumental evaluation to identify if there is an equal or different stiffness between the right and left ileotibial band.
  Interventions: Other: Manual evaluation of ITB tension

INTERVENTIONS:
Other: Manual evaluation of ITB tension — There will be a double evaluation for each sampling session: 1) if there is a uniformity of the tension between the two sides, or if there is a prevalence on one side; 2) quantification of the difference, if present, with a graduation in 3 levels.

SUMMARY:
The goal of this clinical-test study is to evaluate the reliability of the direct palpation of the ileotibial band. For this purpose, a group of 100 healthy subjects will be considered. The main question it aims to answer regards the reproducibility of the intra and inter examiner evaluation performed on the same day (intra-day) and the validation of the palpatory examination with an instrumental measure of the tissue tension.

Participants will undergo a manual and instrumental sampling of the ileotibial band tension of both legs.

DETAILED DESCRIPTION:
The project includes 6 phases:

I phase - agreement in principle on the method of collection; II phase - recruitment; III phase - first sampling; IV phase - training on perception and concordance; V phase - second sampling to verify the progression of the agreement; VI phase - third manual sampling and evaluation with Myoton.

Description of the phases

Phase I - Two examiners together with the principal investigator perform 2 hours of training to standardize the sampling method (localization of the point to be evaluated of the Iileotibial band -ITB- and intensity of pressure of the fingertips to be used) and discussion on the tension gradation detected on the ITB with some volunteers.

Phase II - The recruitment will be carried out through the search for volunteers among the students of the OSCE-Bologna school of osteopathy, through announcement in the classroom and publication of the recruitment in the FB social group of the school (OSCE planet) and WhatsApp groups of students organized by year .

Phase III - First sampling of manual evaluation only, using a sample of 40 subjects (both limbs), as proposed in the literature.

The detection is to identify if there is an equal or different stiffness between the right and left ITB.

The transcript of the discovery will be double for each sampling session: 1) the first will report whether there is a uniformity of the tension between the two sides, or if there is a prevalence on one side; the second will try to quantify, in case there is a difference between the two sides, with a graduation of 3 levels of the difference.

In the first survey, the examiner will indicate a higher tension on the right side with +1; - 1 on the left side; 0 if there are no significant differences.

The second detection is to identify, when present, the graduation of the stiffness difference between the two sides, arbitrarily divided into 3 levels. The examiner, therefore, will report:

* 3 to indicate greater tension on the right with a large difference from the left;
* 2 to indicate a higher tension on the right with an average difference compared to the left;
* 1 to indicate greater tension on the right with a slight difference from the left; 0 to indicate a non-appreciable prevalence of tension on one side over the other;

  * 3 to indicate greater tension on the left with a large difference compared to the right;
  * 2 to indicate a greater tension on the left with an average difference compared to the right;
  * 1 to indicate more tension on the left with a slight difference from the right.

IV phase - The manual examiners carry out a training period on perception and concordance, lasting about 20 hours. This training is carried out using instruments (gold standard) made specifically to modify the state of stiffness of elastic structures and strings that simulate the ITB, connected to dynamometers to measure the amount of stiffness. In vivo evaluation, among the operators, are used to verify the exact positioning where to perform the stiffness sampling and compare the tension data obtained for the construction of the agreement.

V phase - The second sampling to verify the progression of the manual agreement, as proposed in the literature, is carried out by evaluating the stiffness of the ITB, in the same way as for the first sampling with volunteers, but in a reduced sample (about 20 subjects). If the statistical processing of the results of this test evaluation shows a good level in the agreement (Cohen K > 0.60), the definitive sampling is scheduled at a later date; otherwise you return to training by increasing the hours.

VI phase - The definitive manual sampling consists in repeating, using the same method of the first evaluation (baseline), with different or identical subjects of the first sampling. The number of subjects will always be 40, evaluated by both examiners and each examiner will evaluate the same subject twice at a distance of about 20-60 minutes. The same subjects will be tested, after the manual evaluation, with the Myoton using the modality previously described. The Myoton results are automatically stored in the preset instrument with the subject's ID and can be downloaded to the computer in an Excel worksheet.

All the data obtained is collected and processed by the examiner who does not participate directly in the data collection using an Excel spreadsheet and / or the R program.

ELIGIBILITY:
Inclusion Criteria:

- healthy subjects

Exclusion Criteria:

* clinically evident painful symptoms that, in the opinion of the subject himself or the examiner, may prevent the test from being carried out (for example, pain in the hip while maintaining the sampling position);
* evident excess weight (BMI greater than 28 kg / m2) which may make the manual and instrumental result obtained doubtful.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Precision of the palpation test | 5 seconds for each evaluation (day 1)
  intra-day concordance intra and inter examiners by means of weighted Cohen's K with use of sampling evaluation divided into 3 intervals (+1, 0, -1) and 7 intervals (+3, +2, +1, 0, -1, -2, -3)

SECONDARY OUTCOMES:
Effect of training | 5 seconds for each evaluation (day 1)
  Evaluation of how a dedicated training / agreement can modify the level of agreement between intra and inter examiner, by means of weighted Cohen's K with use of sampling evaluation divided into 3 intervals (+1, 0, -1) and 7 intervals (+3, +2, +1, 0, -1, -2, -3)
Accuracy of the palpation test | 5 seconds for each evaluation (day 1)
  Concordance intra-day between the manual and instrument evaluation. The instrumental data are processed by subtracting the average data of the three measurements (automatically carried out by the instrument) of the right limb from that of the left. The data obtained is categorized into 3 levels to be compared, again using weighted Cohen's K, with the data from the manual evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Spine Center, Bologna, Italy

REFERENCES:
- [Background] Arab AM, Nourbakhsh MR. The relationship between hip abductor muscle strength and iliotibial band tightness in individuals with low back pain. Chiropr Osteopat. 2010 Jan 13;18:1. doi: 10.1186/1746-1340-18-1. PMID 20157442
- [Background] Chen G, Wu J, Chen G, Lu Y, Ren W, Xu W, Xu X, Wu Z, Guan Y, Zheng Y, Qiu B. Reliability of a portable device for quantifying tone and stiffness of quadriceps femoris and patellar tendon at different knee flexion angles. PLoS One. 2019 Jul 31;14(7):e0220521. doi: 10.1371/journal.pone.0220521. eCollection 2019. PMID 31365582
- [Background] Cibulka MT, Bennett J. How weakness of the tensor fascia lata and gluteus maximus may contribute to ACL injury: A new theory. Physiother Theory Pract. 2020 Mar;36(3):359-364. doi: 10.1080/09593985.2018.1486492. Epub 2018 Jun 21. PMID 29927670
- [Background] Friede MC, Klauser A, Fink C, Csapo R. Stiffness of the iliotibial band and associated muscles in runner's knee: Assessing the effects of physiotherapy through ultrasound shear wave elastography. Phys Ther Sport. 2020 Sep;45:126-134. doi: 10.1016/j.ptsp.2020.06.015. Epub 2020 Jul 25. PMID 32769015
- [Background] Patijn, J. Reproducibility protocol for diagnostic procedures in Manual/Musculoskeletal Medicine. Manuelle Medizin 2019; 57, 451-479.
- [Background] Melchione WE, Sullivan MS. Reliability of measurements obtained by use of an instrument designed to indirectly measure iliotibial band length. J Orthop Sports Phys Ther. 1993 Sep;18(3):511-5. doi: 10.2519/jospt.1993.18.3.511. PMID 8298633
- [Background] Garcia-Bernal MI, Heredia-Rizo AM, Gonzalez-Garcia P, Cortes-Vega MD, Casuso-Holgado MJ. Validity and reliability of myotonometry for assessing muscle viscoelastic properties in patients with stroke: a systematic review and meta-analysis. Sci Rep. 2021 Mar 3;11(1):5062. doi: 10.1038/s41598-021-84656-1. PMID 33658623

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT05782439/Prot_SAP_000.pdf